CLINICAL TRIAL: NCT00831103
Title: A Randomized, Double-blind, Active-controlled, Multi-center, Parallel-group Dose-ranging Study Assessing the Safety and Efficacy of EPB-348 Versus Valacyclovir Among Immunocompetent Patients With an Acute Episode of Herpes Zoster
Brief Title: A Phase 2b Trial of EPB-348 for the Treatment of Herpes Zoster
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epiphany Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPB348-0201
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Herpes Zoster
Keywords: EPB348; Valomaciclovir Stearate; Valacyclovir; Herpes Zoster; Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- EPB-348 1000 mg (Experimental): EPB-348 1000 mg dosed once daily for seven days
  Interventions: Drug: EPB-348
- EPB-348 2000 mg (Experimental): EPB-348 2000 mg dosed once daily for seven days
  Interventions: Drug: EPB-348
- EPB-348 3000 mg (Experimental): EPB-348 3000 mg dosed once daily for seven days
  Interventions: Drug: EPB-348
- Valacyclovir (Active Comparator): Valacyclovir 1000 mg dosed three times daily for seven days
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: EPB-348 — Treated over seven days
  Other Names: Valomaciclovir Stearate
  Arms: EPB-348 1000 mg; EPB-348 2000 mg; EPB-348 3000 mg
Drug: Valacyclovir — Treated over seven days
  Other Names: Valtrex
  Arms: Valacyclovir

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and dosage of EPB-348 that best balances safety and efficacy among adult immunocompetent patients with an acute episode of herpes zoster.

DETAILED DESCRIPTION:
In cells infected with varicella-zoster virus, there is evidence to suggest that EPB-348 could offer clinically important advantages in the treatment of acute herpes zoster over currently available therapies due to rapid absorption and conversion to the active moiety as well as a longer intra-cellular half-life in infected cells. Clinically, these characteristics could translate into once-daily dosing versus thrice-daily dosing as seen with current therapy, leading to a higher rate of compliance and quality-of-life, especially among elderly patients. The objective of EPB348-0201 is to determine the pharmacokinetics and dosage of EPB-348 that best balances safety and efficacy among adult immunocompetent patients with an acute episode of herpes zoster. This multi-center study will randomly assign patients to either EPB-348 1000 mg once daily or EPB-348 2000 mg once daily or valacyclovir 1000 mg three times daily.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults at least 18 years of age
* Patients with signs and symptoms consistent with acute herpes zoster disease, namely, a dermatomal vesicular rash which may be preceded by pain and parasthesias in the days before vesicular eruption
* Herpes Zoster associated rash present for ≤ 72 hours
* Patients who are deemed to be immunocompetent based on history and physical exam

Exclusion Criteria:

* Females who are pregnant or nursing
* History or clinical manifestations of significant metabolic, hematological, pulmonary, ischemic, or unstable heart disease, gastrointestinal, neurological, psychiatric, renal, urological, endocrine, opthalmologic, or immune mediated disease including HIV or HBsAg positivity
* Chronic genital herpes
* Patients who received cytotoxic or immunosuppressive drug therapy within 3 months prior to study participation
* Previous vaccinations against Herpes Zoster
* Patients with > 50% of vesicles crusted at screen
* Patients who received topical or systemic antiviral medications or immunomodulatory agents for herpes zoster viral infections or capsaicin within 4 weeks of study participation
* Patients with a history of congenital, acquired, or corticosteroid induced immunodeficiency, including malignancy, significantly impaired renal function (creatinine clearance < 50 cc/min), and impaired hepatic function (ALT or AST levels > 3 times the upper limit of normal)
* QTc > 500msec
* Patients with a history of intolerance or hypersensitivity to acyclovir, penciclovir, valacyclovir, or famciclovir
* Patients with gastrointestinal dysfunction that might interfere with drug absorption
* Patients, considered by the investigator, for any reason, to be an unsuitable candidate for receiving the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To compare the time-to-crusting of vesicles on patients in each of the EPB-348 dosing arms versus the valacyclovir dosing arm. | Daily assessment during the seven days of treament then weekly until Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K Tyring, MD, Principal Investigator — University of Texas Health Science Center, Houston, Texas
Locations (1):
- Center for Clinical Studies-Medical Center, Houston, Texas, United States

REFERENCES:
- [Result] Tyring SK, Plunkett S, Scribner AR, Broker RE, Herrod JN, Handke LT, Wise JM, Martin PA; Valomaciclovir Zoster Study Group. Valomaciclovir versus valacyclovir for the treatment of acute herpes zoster in immunocompetent adults: a randomized, double-blind, active-controlled trial. J Med Virol. 2012 Aug;84(8):1224-32. doi: 10.1002/jmv.23329. PMID 22711350